CLINICAL TRIAL: NCT00315926
Title: Melatonin and Cardiac Morbidity After Elective Abdominal Aortic Aneurism Repair
Brief Title: Melatonin and Cardiac Outcome After Major Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Dr. Bülent Kücükakin, dept. of surgery, Gentofte Hospital, Copenhagen, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2612-3109
Record Dates: First submitted 2006-04-18; First posted 2006-04-19 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2006-11

CONDITIONS: Aortic Aneurysm
Keywords: Cardiac morbidity; Melatonin; Surgery; Postoperative
MeSH Terms: conditions — Aortic Aneurysm | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin (Experimental)
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — Melatonin 50 mg during surgery and 10 mg every night for 3 nights
  Arms: Melatonin
Drug: Placebo — a mixture of ethanol and physiological saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess whether treatment with melatonin can reduce cell damage and inflammatory stress response and thereby occurrence of myocardial injury after abdominal aortic surgery.

DETAILED DESCRIPTION:
Abdominal aortic surgery is associated with a significant increase of oxidative and inflammatory stress response. Aortic surgery is also associated with elevated troponin which is a sensitive and specific marker for myocardial injury. The severity of oxidative stress is correlated with elevated troponin. Melatonin, which is a hormone produced in brain, seems to modify cell damage and inflammation. On the other hand we know, that melatonin production first night after surgery is disturbed. The purpose of this study is therefore to determine whether treatment with melatonin can reduce cell damage and inflammation, and thereby occurrence of myocardial injury associated with abdominal aortic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Indication for elective abdominal aortic aneurism surgery or periphery atheroscleroses with indicated protheses operation
* Patients between 18 and 80 years old

Exclusion Criteria:

* Patients with ASA class > 3
* Anticoagulation therapy (marevan and marcoumar)
* Preoperative therapy with opioid, anxiolytic and hypnotic medication
* Renal insufficient (preoperative creatinin > 200 mmol/l)
* Well-known liver insufficient
* Alcohol consumption (more than 5 drinks)
* Compliance (language difficulty, mental problems etc.)
* Pregnancy and breast-feeding
* Lack of written consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Cardiac morbidity | 30 days
  artrial fibrillation, unstable angina, myocardial infarction, ECG changes (T-wave inversion for more than 24 hours, new ST-segment depression for more than 24 hours, acute ST-segment elevation with appearance of q-waves or loss of R-waves, left bundle branch block), or a characteristic pattern of rising and falling values of troponin-I, or pulmonary oedema. Mortality was defined as any cause of death in the 30 days after surgery.

SECONDARY OUTCOMES:
Oxidative and inflammatory stress response | 3 days
  Blood samples for analysis of malondialdehyde (MDA), ascorbic acid (AA), dehydroascorbic acid (DHA) and C-reactive protein (CRP) assessed before and after operation

CONTACTS AND LOCATIONS:
Overall Officials: Bülent Kücükakin, Principal Investigator — Department of Surgical Gastroenterology, University Hospital of Copenhagen in Gentofte
Locations (1):
- Department of Surgical Gastroenterology, University Hospital of Copenhagen in Gentofte, Hellerup, Denmark